CLINICAL TRIAL: NCT07322458
Title: The Effect of Spinal Cord Stimulation on Orthostatic Hypotension in Parkinsonism and Its Related Mechanisms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDS_OH_tSCS
Record Dates: First submitted 2025-12-21; First posted 2026-01-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-09

CONDITIONS: Parkinsonism
MeSH Terms: conditions — Parkinsonian Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural spinal cord stimulation (eSCS) implantation (Experimental): Phase I: (1) Spinal cord segment is selected as the puncture location according to the patient's symptom and the condition of the patient's spinal cord. Percutaneous puncture is performed under X-ray guidance. One or two electrodes are placed in the patient's epidural cavity, and the electrode position is adjusted intraoperatively and by the patient's feedback of the current stimulation position until the current can cover the entire area. (2) An extension lead is connected, an external temporary stimulator is attached, and the patient decides whether to proceed to full implantation in phase II after 7-10 days of phase I testing experience. Phase II: The complete SCS system is implanted under local anesthesia or epidural anesthesia after successful testing. A subcutaneous capsular bag is usually created in the lower abdomen and the implanted electrodes are connected to the pulse generator through a connecting wire in the subcutaneous tunnel.
  Interventions: Device: Epidural spinal cord stimulation
- Transcutaneous spinal cord stimulation (tSCS) application (Experimental): After completing the necessary assessments and informed consent procedures, subjects will undergo device installation and seated programming. The cathode of the tSCS device will be placed at the level of the lower thoracic spinal cord via a hydrogel adhesive electrode, and the anode will be placed bilaterally at the iliac crest via a hydrogel adhesive electrode. During seated programming, subjects will undergo continuous non-invasive blood pressure monitoring and a medication-free head-up tilt test (TTT). If subjects demonstrate a satisfactory clinical response during the testing phase (defined as an increase in systolic blood pressure of more than 15-20 mmHg with stimulation on compared to the off state), they will enter regular tSCS therapy during the treatment phase.
  Interventions: Device: Transcutaneous spinal cord stimulation

INTERVENTIONS:
Device: Epidural spinal cord stimulation — Epidural spinal cord stimulation (eSCS) is a very thin electrode implanted in the dorsal epidural space of the spinal cord to improve the patient's symptoms by stimulating the spinal nerves with pulsed electrical currents, which attenuate or enhance the flow of nerve impulses from the periphery to the central system, i.e., stimulating thick fibres to achieve therapeutic results. SCS system consists of three components: an electrode implanted in the epidural space of the patient's spinal cord, a stimulator implanted subcutaneously in the abdomen or buttocks that delivers electrical impulses, and an extension cord that connects the two.
  Arms: Epidural spinal cord stimulation (eSCS) implantation
Device: Transcutaneous spinal cord stimulation — Transcutaneous spinal cord stimulation (tSCS) is a non-invasive treatment that improves symptoms by stimulating spinal nerves with pulsed electrical currents via electrodes placed at corresponding spinal cord segments. The tSCS system consists of an electrical pulse stimulator, wires, and conductive patches.
  Arms: Transcutaneous spinal cord stimulation (tSCS) application

SUMMARY:
Parkinson's disease (PDS) is a syndrome characterized by tremor, bradykinesia, rigidity, and postural disturbances. Causes include Parkinson's disease (PD), multiple system atrophy (MSA), progressive supranuclear palsy (PSP), and corticobasal degeneration (CBD). Non-motor symptoms of PDS, such as neurogenic orthostatic hypotension (nOH), have received more intensive research due to their greater disabling potential compared to motor symptoms. In patients with PD and MSA, nOH can lead to intolerance to medications such as levodopa, significantly increasing the risk of falls, accelerating cognitive decline, and increasing the risk of all-cause mortality. However, conventional pharmacological treatments (such as midodrine, droxidopa, and fludrocortisone) and non-pharmacological approaches (such as compression abdominal bands, elastic stockings, and deep brain stimulation) for non-motor symptoms such as nOH have numerous limitations, including short-term efficacy, uncertain efficacy, and side effects. Therefore, exploring new non-pharmacological treatments to improve nOH and delay disease progression in patients with PDS is crucial for improving their quality of life and prognosis.

Spinal cord stimulation (SCS), including invasive (epidural) spinal cord stimulation (eSCS) and non-invasive (transcutaneous) spinal cord stimulation (tSCS), is a novel neuromodulatory technique with clinical applications in a variety of neurological diseases. Currently, several small-sample studies have suggested the potential efficacy of SCS for nOH caused by spinal cord injury (SCI). This study innovatively proposes the use of eSCS and tSCS to improve nOH and related clinical symptoms in patients with PDS. A prospective, single-center, randomized, controlled clinical trial is planned to compare the efficacy of invasive and non-invasive SCS in treating nOH, thereby providing new insights for the effective treatment of PDS.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged between 40 and 80 years;
* 2. No dementia as measured by the cMMSE scale (formal cMMSE score should be >20 for subjects with 1 to 6 years of formal education; cMMSE score should be >24 for subjects with >6 years of formal education);
* 3. Able and willing to follow instruction of the researcher;
* 4. No other conditions that the researchers consider inappropriate for inclusion:

Exclusion Criteria:

* 1. Severe depression (HAMD-17 above 17 as moderate to severe) or anxiety;
* 2. Pregnancy;
* 3. History of alcoholism;
* 4. No skin abnormalities;
* 5. Non-neurological disease-related symptoms that prevent patients from participation in the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of blood pressure from baseline to immediately post-operation or post transcutaneous stimulation | Immediately post surgery or post transcutaneous stimulation
  Changes of on-off delta systolic and delta diastolic blood pressure from baseline to immediately post-operation or post-stimulation. Delta systolic blood pressure equals the systolic blood pressure of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes. Delta diastolic blood pressure equals the diastolic blood pressure of the patient lying minus the diastolic blood pressure of the patient standing up for 10 minutes.
Change of blood pressure from baseline to 3 months post-operation or post transcutaneous stimulation | 3 months post surgery or post transcutaneous stimulation
  Changes of on-off delta systolic and delta diastolic blood pressure from baseline to 3 months post-operation or post-stimulation. Delta systolic blood pressure equals the systolic blood pressure of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes. Delta diastolic blood pressure equals the diastolic blood pressure of the patient lying minus the diastolic blood pressure of the patient standing up for 10 minutes.
Change of blood pressure from baseline to 6 months post-operation or post transcutaneous stimulation | 6 months post surgery or post transcutaneous stimulation
  Changes of on-off delta systolic and delta diastolic blood pressure from baseline to 6 months post-operation or post-stimulation. Delta systolic blood pressure equals the systolic blood pressure of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes. Delta diastolic blood pressure equals the diastolic blood pressure of the patient lying minus the diastolic blood pressure of the patient standing up for 10 minutes.
Change of blood pressure from baseline to 9 months post-operation or post transcutaneous stimulation | 9 months post surgery or post transcutaneous stimulation
  Changes of on-off delta systolic and delta diastolic blood pressure from baseline to immediately post-operation or post-stimulation. Delta systolic blood pressure equals the systolic blood pressure of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes. Delta diastolic blood pressure equals the diastolic blood pressure of the patient lying minus the diastolic blood pressure of the patient standing up for 10 minutes.
Change of blood pressure from baseline to 12 months post-operation or post transcutaneous stimulation | 12 months post surgery or post transcutaneous stimulation
  Changes of on-off delta systolic and delta diastolic blood pressure from baseline to 12 months post-operation or post-stimulation. Delta systolic blood pressure equals the systolic blood pressure of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes. Delta diastolic blood pressure equals the diastolic blood pressure of the patient lying minus the diastolic blood pressure of the patient standing up for 10 minutes.
Change of blood pressure from baseline to 18 months post-operation or post transcutaneous stimulation | 18 months post surgery or post transcutaneous stimulation
  Changes of on-off delta systolic and delta diastolic blood pressure from baseline to 18 months post-operation or post-stimulation. Delta systolic blood pressure equals the systolic blood pressure of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes. Delta diastolic blood pressure equals the diastolic blood pressure of the patient lying minus the diastolic blood pressure of the patient standing up for 10 minutes.
Change of blood pressure from baseline to 24 months post-operation or post transcutaneous stimulation | 24 months post surgery or post transcutaneous stimulation
  Changes of on-off delta systolic and delta diastolic blood pressure from baseline to 24 months post-operation or post-stimulation. Delta systolic blood pressure equals the systolic blood pressure of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes. Delta diastolic blood pressure equals the diastolic blood pressure of the patient lying minus the diastolic blood pressure of the patient standing up for 10 minutes.

SECONDARY OUTCOMES:
Change of oxygen desaturation index from baseline to immediately post-operation or post transcutaneous stimulation | Immediately post surgery or post transcutaneous stimulation
  Change of oxygen desaturation index measured by on-off polysomnography from baseline to immediately post-operation or post transcutaneous stimulation
Change of oxygen desaturation index from baseline to 3 months post-operation or post transcutaneous stimulation | 3 months post surgery or post transcutaneous stimulation
  Change of oxygen desaturation index measured by on-off polysomnography from baseline to 3 months post-operation or post transcutaneous stimulation
Change of oxygen desaturation index from baseline to 6 months post-operation or post transcutaneous stimulation | 6 months post surgery or post transcutaneous stimulation
  Change of oxygen desaturation index measured by on-off polysomnography from baseline to 6 months post-operation or post transcutaneous stimulation
Change of oxygen desaturation index from baseline to 9 months post-operation or post transcutaneous stimulation | 9 months post surgery or post transcutaneous stimulation
  Change of oxygen desaturation index measured by on-off polysomnography from baseline to 9 months post-operation or post transcutaneous stimulation
Change of oxygen desaturation index from baseline to 12 months post-operation or post transcutaneous stimulation | 12 months post surgery or post transcutaneous stimulation
  Change of oxygen desaturation index measured by on-off polysomnography from baseline to 12 months post-operation or post transcutaneous stimulation
Change of oxygen desaturation index from baseline to 18 months post-operation or post transcutaneous stimulation | 18 months post surgery or post transcutaneous stimulation
  Change of oxygen desaturation index measured by on-off polysomnography from baseline to 18 months post-operation or post transcutaneous stimulation
Change of oxygen desaturation index from baseline to 24 months post-operation or post transcutaneous stimulation | 24 months post surgery or post transcutaneous stimulation
  Change of oxygen desaturation index measured by on-off polysomnography from baseline to 24 months post-operation or post transcutaneous stimulation
Change of apnea hypopnea index from baseline to immediately post-operation or post transcutaneous stimulation | Immediately post surgery or post transcutaneous stimulation
  Change of apnea hypopnea index measured by on-off polysomnography from baseline to immediately post-operation or post transcutaneous stimulation
Change of apnea hypopnea index from baseline to 3 months post-operation or post transcutaneous stimulation | 3 months post surgery or post transcutaneous stimulation
  Change of apnea hypopnea index measured by on-off polysomnography from baseline to 3 months post-operation or post transcutaneous stimulation
Change of apnea hypopnea index from baseline to 6 months post-operation or post transcutaneous stimulation | 6 months post surgery or post transcutaneous stimulation
  Change of apnea hypopnea index measured by on-off polysomnography from baseline to 6 months post-operation or post transcutaneous stimulation
Change of apnea hypopnea index from baseline to 9 months post-operation or post transcutaneous stimulation | 9 months post surgery or post transcutaneous stimulation
  Change of apnea hypopnea index measured by on-off polysomnography from baseline to 9 months post-operation or post transcutaneous stimulation
Change of apnea hypopnea index from baseline to 12 months post-operation or post transcutaneous stimulation | 12 months post surgery or post transcutaneous stimulation
  Change of apnea hypopnea index measured by on-off polysomnography from baseline to 12 months post-operation or post transcutaneous stimulation
Change of apnea hypopnea index from baseline to 18 months post-operation or post transcutaneous stimulation | 18 months post surgery or post transcutaneous stimulation
  Change of apnea hypopnea index measured by on-off polysomnography from baseline to 18 months post-operation or post transcutaneous stimulation
Change of apnea hypopnea index from baseline to 24 months post-operation or post transcutaneous stimulation | 24 months post surgery or post transcutaneous stimulation
  Change of apnea hypopnea index measured by on-off polysomnography from baseline to 24 months post-operation or post transcutaneous stimulation
Change of on-off 24-hour blood pressure monitoring from baseline to immediately post-operation or post transcutaneous stimulation | Immediately post surgery or post transcutaneous stimulation
  Change of on-off 24-hour blood pressure monitoring from baseline to immediately post-operation or post transcutaneous stimulation
Change of on-off 24-hour blood pressure monitoring from baseline to 3 months post-operation or post transcutaneous stimulation | 3 months post surgery or post transcutaneous stimulation
  Change of on-off 24-hour blood pressure monitoring from baseline to 3 months post-operation or post transcutaneous stimulation
Change of on-off 24-hour blood pressure monitoring from baseline to 6 months post-operation or post transcutaneous stimulation | 6 months post surgery or post transcutaneous stimulation
  Change of on-off 24-hour blood pressure monitoring from baseline to 6 months post-operation or post transcutaneous stimulation
Change of on-off 24-hour blood pressure monitoring from baseline to 9 months post-operation or post transcutaneous stimulation | 9 months post surgery or post transcutaneous stimulation
  Change of on-off 24-hour blood pressure monitoring from baseline to 9 months post-operation or post transcutaneous stimulation
Change of on-off 24-hour blood pressure monitoring from baseline to 12 months post-operation or post transcutaneous stimulation | 12 months post surgery or post transcutaneous stimulation
  Change of on-off 24-hour blood pressure monitoring from baseline to 12 months post-operation or post transcutaneous stimulation
Change of on-off 24-hour blood pressure monitoring from baseline to 18 months post-operation or post transcutaneous stimulation | 18 months post surgery or post transcutaneous stimulation
  Change of on-off 24-hour blood pressure monitoring from baseline to 18 months post-operation or post transcutaneous stimulation
Change of on-off 24-hour blood pressure monitoring from baseline to 24 months post-operation or post transcutaneous stimulation | 24 months post surgery or post transcutaneous stimulation
  Change of on-off 24-hour blood pressure monitoring from baseline to 24 months post-operation or post transcutaneous stimulation
Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to immediately post-operation or post transcutaneous stimulation | Immediately post surgery or post transcutaneous stimulation
  Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to immediately post-operation or post transcutaneous stimulation
Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 3 months post-operation or post transcutaneous stimulation | 3 months post surgery or post transcutaneous stimulation
  Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 3 months post-operation or post transcutaneous stimulation
Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 6 months post-operation or post transcutaneous stimulation | 6 months post surgery or post transcutaneous stimulation
  Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 6 months post-operation or post transcutaneous stimulation
Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 9 months post-operation or post transcutaneous stimulation | 9 months post surgery or post transcutaneous stimulation
  Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 9 months post-operation or post transcutaneous stimulation
Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 12 months post-operation or post transcutaneous stimulation | 12 months post surgery or post transcutaneous stimulation
  Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 12 months post-operation or post transcutaneous stimulation
Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 18 months post-operation or post transcutaneous stimulation | 18 months post surgery or post transcutaneous stimulation
  Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 18 months post-operation or post transcutaneous stimulation
Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 24 months post-operation or post transcutaneous stimulation | 24 months post surgery or post transcutaneous stimulation
  Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 24 months post-operation or post transcutaneous stimulation
Change of serum catecholamine neurotransmitter levels from baseline to immediately post-operation or post transcutaneous stimulation | Immediately post surgery or post transcutaneous stimulation
  Change of on-off delta serum catecholamine neurotransmitter levels from baseline to immediately post-operation or post transcutaneous stimulation. Delta serum catecholamine neurotransmitter levels equals the serum catecholamine neurotransmitter levels of the patient lying minus the serum catecholamine neurotransmitter levels of the patient standing up for 10 minutes.
Change of serum catecholamine neurotransmitter levels from baseline to 3 months post-operation or post transcutaneous stimulation | 3 months post surgery or post transcutaneous stimulation
  Change of on-off delta serum catecholamine neurotransmitter levels from baseline to 3 months post-operation or post transcutaneous stimulation. Delta serum catecholamine neurotransmitter levels equals the serum catecholamine neurotransmitter levels of the patient lying minus the serum catecholamine neurotransmitter levels of the patient standing up for 10 minutes.
Change of serum catecholamine neurotransmitter levels from baseline to 6 months post-operation or post transcutaneous stimulation | 6 months post surgery or post transcutaneous stimulation
  Change of on-off delta serum catecholamine neurotransmitter levels from baseline to 6 months post-operation or post transcutaneous stimulation. Delta serum catecholamine neurotransmitter levels equals the serum catecholamine neurotransmitter levels of the patient lying minus the serum catecholamine neurotransmitter levels of the patient standing up for 10 minutes.
Change of serum catecholamine neurotransmitter levels from baseline to 9 months post-operation or post transcutaneous stimulation | 9 months post surgery or post transcutaneous stimulation
  Change of on-off delta serum catecholamine neurotransmitter levels from baseline to 9 months post-operation or post transcutaneous stimulation. Delta serum catecholamine neurotransmitter levels equals the serum catecholamine neurotransmitter levels of the patient lying minus the serum catecholamine neurotransmitter levels of the patient standing up for 10 minutes.
Change of serum catecholamine neurotransmitter levels from baseline to 12 months post-operation or post transcutaneous stimulation | 12 months post surgery or post transcutaneous stimulation
  Change of on-off delta serum catecholamine neurotransmitter levels from baseline to 12 months post-operation or post transcutaneous stimulation. Delta serum catecholamine neurotransmitter levels equals the serum catecholamine neurotransmitter levels of the patient lying minus the serum catecholamine neurotransmitter levels of the patient standing up for 10 minutes.
Change of serum catecholamine neurotransmitter levels from baseline to 18 months post-operation or post transcutaneous stimulation | 18 months post surgery or post transcutaneous stimulation
  Change of on-off delta serum catecholamine neurotransmitter levels from baseline to 18 months post-operation or post transcutaneous stimulation. Delta serum catecholamine neurotransmitter levels equals the serum catecholamine neurotransmitter levels of the patient lying minus the serum catecholamine neurotransmitter levels of the patient standing up for 10 minutes.
Change of serum catecholamine neurotransmitter levels from baseline to 24 months post-operation or post transcutaneous stimulation | 24 months post surgery or post transcutaneous stimulation
  Change of on-off delta serum catecholamine neurotransmitter levels from baseline to 24 months post-operation or post transcutaneous stimulation. Delta serum catecholamine neurotransmitter levels equals the serum catecholamine neurotransmitter levels of the patient lying minus the serum catecholamine neurotransmitter levels of the patient standing up for 10 minutes.
Change of on-off delta heart rate variability from baseline to immediately post-operation or post transcutaneous stimulation | Immediately post surgery or post transcutaneous stimulation
  Change of on-off delta heart rate variability from baseline to immediately post-operation or post transcutaneous stimulation. Delta heart rate variability equals the heart rate variability of the patient lying minus the heart rate variability of the patient standing up for 10 minutes.
Change of on-off delta heart rate variability from baseline to 3 months post-operation or post transcutaneous stimulation | 3 months post surgery or post transcutaneous stimulation
  Change of on-off delta heart rate variability from baseline to 3 months post-operation or post transcutaneous stimulation. Delta heart rate variability equals the heart rate variability of the patient lying minus the heart rate variability of the patient standing up for 10 minutes.
Change of on-off delta heart rate variability from baseline to 6 months post-operation or post transcutaneous stimulation | 6 months post surgery or post transcutaneous stimulation
  Change of on-off delta heart rate variability from baseline to 6 months post-operation or post transcutaneous stimulation. Delta heart rate variability equals the heart rate variability of the patient lying minus the heart rate variability of the patient standing up for 10 minutes.
Change of on-off delta heart rate variability from baseline to 9 months post-operation or post transcutaneous stimulation | 9 months post surgery or post transcutaneous stimulation
  Change of on-off delta heart rate variability from baseline to 9 months post-operation or post transcutaneous stimulation. Delta heart rate variability equals the heart rate variability of the patient lying minus the heart rate variability of the patient standing up for 10 minutes.
Change of on-off delta heart rate variability from baseline to 12 months post-operation or post transcutaneous stimulation | 12 months post surgery or post transcutaneous stimulation
  Change of on-off delta heart rate variability from baseline to 12 months post-operation or post transcutaneous stimulation. Delta heart rate variability equals the heart rate variability of the patient lying minus the heart rate variability of the patient standing up for 10 minutes.
Change of on-off delta heart rate variability from baseline to 18 months post-operation or post transcutaneous stimulation | 18 months post surgery or post transcutaneous stimulation
  Change of on-off delta heart rate variability from baseline to 18 months post-operation or post transcutaneous stimulation. Delta heart rate variability equals the heart rate variability of the patient lying minus the heart rate variability of the patient standing up for 10 minutes.
Change of on-off delta heart rate variability from baseline to 24 months post-operation or post transcutaneous stimulation | 24 months post surgery or post transcutaneous stimulation
  Change of on-off delta heart rate variability from baseline to 24 months post-operation or post transcutaneous stimulation. Delta heart rate variability equals the heart rate variability of the patient lying minus the heart rate variability of the patient standing up for 10 minutes.
Change of length of walking during 6-minute walking test from baseline to immediately post-operation or post transcutaneous stimulation | Immediately post surgery or post transcutaneous stimulation
  Change of on-off length of walking during 6-minute walking test from baseline to immediately post-operation or post transcutaneous stimulation
Change of length of walking during 6-minute walking test from baseline to 3 months post-operation or post transcutaneous stimulation | 3 months post surgery or post transcutaneous stimulation
  Change of on-off length of walking during 6-minute walking test from baseline to 3 months post-operation or post transcutaneous stimulation
Change of length of walking during 6-minute walking test from baseline to 6 months post-operation or post transcutaneous stimulation | 6 months post surgery or post transcutaneous stimulation
  Change of on-off length of walking during 6-minute walking test from baseline to 6 months post-operation or post transcutaneous stimulation
Change of length of walking during 6-minute walking test from baseline to 9 months post-operation or post transcutaneous stimulation | 9 months post surgery or post transcutaneous stimulation
  Change of on-off length of walking during 6-minute walking test from baseline to 9 months post-operation or post transcutaneous stimulation
Change of length of walking during 6-minute walking test from baseline to 12 months post-operation or post transcutaneous stimulation | 12 months post surgery or post transcutaneous stimulation
  Change of on-off length of walking during 6-minute walking test from baseline to 12 months post-operation or post transcutaneous stimulation
Change of length of walking during 6-minute walking test from baseline to 18 months post-operation or post transcutaneous stimulation | 18 months post surgery or post transcutaneous stimulation
  Change of on-off length of walking during 6-minute walking test from baseline to 18 months post-operation or post transcutaneous stimulation
Change of length of walking during 6-minute walking test from baseline to 24 months post-operation or post transcutaneous stimulation | 24 months post surgery or post transcutaneous stimulation
  Change of on-off length of walking during 6-minute walking test from baseline to 24 months post-operation or post transcutaneous stimulation
Change of time of walking during 6-minute walking test from baseline to immediately post-operation or post transcutaneous stimulation | Immediately post surgery or post transcutaneous stimulation
  Change of on-off time of walking during 6-minute walking test from baseline to immediately post-operation or post transcutaneous stimulation
Change of time of walking during 6-minute walking test from baseline to 3 months post-operation or post transcutaneous stimulation | 3 months post surgery or post transcutaneous stimulation
  Change of on-off time of walking during 6-minute walking test from baseline to 3 months post-operation or post transcutaneous stimulation
Change of time of walking during 6-minute walking test from baseline to 6 months post-operation or post transcutaneous stimulation | 6 months post surgery or post transcutaneous stimulation
  Change of on-off time of walking during 6-minute walking test from baseline to 6 months post-operation or post transcutaneous stimulation
Change of time of walking during 6-minute walking test from baseline to 9 months post-operation or post transcutaneous stimulation | 9 months post surgery or post transcutaneous stimulation
  Change of on-off time of walking during 6-minute walking test from baseline to 9 months post-operation or post transcutaneous stimulation
Change of time of walking during 6-minute walking test from baseline to 12 months post-operation or post transcutaneous stimulation | 12 months post surgery or post transcutaneous stimulation
  Change of on-off time of walking during 6-minute walking test from baseline to 12 months post-operation or post transcutaneous stimulation
Change of time of walking during 6-minute walking test from baseline to 18 months post-operation or post transcutaneous stimulation | 18 months post surgery or post transcutaneous stimulation
  Change of on-off time of walking during 6-minute walking test from baseline to 18 months post-operation or post transcutaneous stimulation
Change of time of walking during 6-minute walking test from baseline to 24 months post-operation or post transcutaneous stimulation | 24 months post surgery or post transcutaneous stimulation
  Change of on-off time of walking during 6-minute walking test from baseline to 24 months post-operation or post transcutaneous stimulation
Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to immediately post-operation or post transcutaneous stimulation | Immediately post surgery or post transcutaneous stimulation
  Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to immediately post-operation or post transcutaneous stimulation
Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 3 months post-operation or post transcutaneous stimulation | 3 months post surgery or post transcutaneous stimulation
  Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 3 months post-operation or post transcutaneous stimulation
Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 6 months post-operation or post transcutaneous stimulation | 6 months post surgery or post transcutaneous stimulation
  Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 6 months post-operation or post transcutaneous stimulation
Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 9 months post-operation or post transcutaneous stimulation | 9 months post surgery or post transcutaneous stimulation
  Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 9 months post-operation or post transcutaneous stimulation
Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 12 months post-operation or post transcutaneous stimulation | 12 months post surgery or post transcutaneous stimulation
  Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 12 months post-operation or post transcutaneous stimulation
Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 18 months post-operation or post transcutaneous stimulation | 18 months post surgery or post transcutaneous stimulation
  Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 18 months post-operation or post transcutaneous stimulation
Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 24 months post-operation or post transcutaneous stimulation | 24 months post surgery or post transcutaneous stimulation
  Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 24 months post-operation or post transcutaneous stimulation
Change of on-off time to complete the Stroop Color and Word Test from baseline to immediately post-operation or post transcutaneous stimulation | Immediately post surgery or post transcutaneous stimulation
  Change of on-off time to complete the Stroop Color and Word Test from baseline to immediately post-operation or post transcutaneous stimulation
Change of on-off time to complete the Stroop Color and Word Test from baseline to 3 months post-operation or post transcutaneous stimulation | 3 months post surgery or post transcutaneous stimulation
  Change of on-off time to complete the Stroop Color and Word Test from baseline to 3 months post-operation or post transcutaneous stimulation
Change of on-off time to complete the Stroop Color and Word Test from baseline to 6 months post-operation or post transcutaneous stimulation | 6 months post surgery or post transcutaneous stimulation
  Change of on-off time to complete the Stroop Color and Word Test from baseline to 6 months post-operation or post transcutaneous stimulation
Change of on-off time to complete the Stroop Color and Word Test from baseline to 9 months post-operation or post transcutaneous stimulation | 9 months post surgery or post transcutaneous stimulation
  Change of on-off time to complete the Stroop Color and Word Test from baseline to 9 months post-operation or post transcutaneous stimulation
Change of on-off time to complete the Stroop Color and Word Test from baseline to 12 months post-operation or post transcutaneous stimulation | 12 months post surgery or post transcutaneous stimulation
  Change of on-off time to complete the Stroop Color and Word Test from baseline to 12 months post-operation or post transcutaneous stimulation
Change of on-off time to complete the Stroop Color and Word Test from baseline to 18 months post-operation or post transcutaneous stimulation | 18 months post surgery or post transcutaneous stimulation
  Change of on-off time to complete the Stroop Color and Word Test from baseline to 18 months post-operation or post transcutaneous stimulation
Change of on-off time to complete the Stroop Color and Word Test from baseline to 24 months post-operation or post transcutaneous stimulation | 24 months post surgery or post transcutaneous stimulation
  Change of on-off time to complete the Stroop Color and Word Test from baseline to 24 months post-operation or post transcutaneous stimulation
Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to immediately post-operation or post transcutaneous stimulation | Immediately post surgery or post transcutaneous stimulation
  Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to immediately post-operation or post transcutaneous stimulation. Delta brain cortex oxygenated hemoglobin levels equals the brain cortex oxygenated hemoglobin levels of the patient lying minus the brain cortex oxygenated hemoglobin levels of the patient standing up for 10 minutes.
Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 3 months post-operation or post transcutaneous stimulation | 3 months post surgery or post transcutaneous stimulation
  Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 3 months post-operation or post transcutaneous stimulation. Delta brain cortex oxygenated hemoglobin levels equals the brain cortex oxygenated hemoglobin levels of the patient lying minus the brain cortex oxygenated hemoglobin levels of the patient standing up for 10 minutes.
Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 6 months post-operation or post transcutaneous stimulation | 6 months post surgery or post transcutaneous stimulation
  Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 6 months post-operation or post transcutaneous stimulation. Delta brain cortex oxygenated hemoglobin levels equals the brain cortex oxygenated hemoglobin levels of the patient lying minus the brain cortex oxygenated hemoglobin levels of the patient standing up for 10 minutes.
Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 9 months post-operation or post transcutaneous stimulation | 9 months post surgery or post transcutaneous stimulation
  Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 9 months post-operation or post transcutaneous stimulation. Delta brain cortex oxygenated hemoglobin levels equals the brain cortex oxygenated hemoglobin levels of the patient lying minus the brain cortex oxygenated hemoglobin levels of the patient standing up for 10 minutes.
Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 12 months post-operation or post transcutaneous stimulation | 12 months post surgery or post transcutaneous stimulation
  Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 12 months post-operation or post transcutaneous stimulation. Delta brain cortex oxygenated hemoglobin levels equals the brain cortex oxygenated hemoglobin levels of the patient lying minus the brain cortex oxygenated hemoglobin levels of the patient standing up for 10 minutes.
Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 18 months post-operation or post transcutaneous stimulation | 18 months post surgery or post transcutaneous stimulation
  Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 18 months post-operation or post transcutaneous stimulation. Delta brain cortex oxygenated hemoglobin levels equals the brain cortex oxygenated hemoglobin levels of the patient lying minus the brain cortex oxygenated hemoglobin levels of the patient standing up for 10 minutes.
Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 24 months post-operation or post transcutaneous stimulation | 24 months post surgery or post transcutaneous stimulation
  Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 24 months post-operation or post transcutaneous stimulation. Delta brain cortex oxygenated hemoglobin levels equals the brain cortex oxygenated hemoglobin levels of the patient lying minus the brain cortex oxygenated hemoglobin levels of the patient standing up for 10 minutes.
Change of dysarthria symptom from baseline to immediately post-operation or post transcutaneous stimulation | Immediately post surgery or post transcutaneous stimulation
  Change of dysarthria symptom measured by on-off Dysphonia Severity Index of Atoms Speech Assessment System from baseline to immediately post-operation or post transcutaneous stimulation
Change of dysarthria symptom from baseline to 3 months post-operation or post transcutaneous stimulation | 3 months post surgery or post transcutaneous stimulation
  Change of dysarthria symptom measured by on-off Dysphonia Severity Index of Atoms Speech Assessment System from baseline to 3 months post-operation or post transcutaneous stimulation
Change of dysarthria symptom from baseline to 6 months post-operation or post transcutaneous stimulation | 6 months post surgery or post transcutaneous stimulation
  Change of dysarthria symptom measured by on-off Dysphonia Severity Index of Atoms Speech Assessment System from baseline to 6 months post-operation or post transcutaneous stimulation
Change of dysarthria symptom from baseline to 9 months post-operation or post transcutaneous stimulation | 9 months post surgery or post transcutaneous stimulation
  Change of dysarthria symptom measured by on-off Dysphonia Severity Index of Atoms Speech Assessment System from baseline to 9 months post-operation or post transcutaneous stimulation
Change of dysarthria symptom from baseline to 12 months post-operation or post transcutaneous stimulation | 12 months post surgery or post transcutaneous stimulation
  Change of dysarthria symptom measured by on-off Dysphonia Severity Index of Atoms Speech Assessment System from baseline to 12 months post-operation or post transcutaneous stimulation
Change of dysarthria symptom from baseline to 18 months post-operation or post transcutaneous stimulation | 18 months post surgery or post transcutaneous stimulation
  Change of dysarthria symptom measured by on-off Dysphonia Severity Index of Atoms Speech Assessment System from baseline to 18 months post-operation or post transcutaneous stimulation
Change of dysarthria symptom from baseline to 24 months post-operation or post transcutaneous stimulation | 24 months post surgery or post transcutaneous stimulation
  Change of dysarthria symptom measured by on-off Dysphonia Severity Index of Atoms Speech Assessment System from baseline to 24 months post-operation or post transcutaneous stimulation
Change of urinary retention from baseline to immediately post-operation or post transcutaneous stimulation | Immediately post surgery or post transcutaneous stimulation
  The change of volume of urinary retention measured by ultrasound and urodynamic study from baseline to immediately post-operation or post transcutaneous stimulation
Change of urinary retention from baseline to 3 months post-operation or post transcutaneous stimulation | 3 months post surgery or post transcutaneous stimulation
  The change of volume of urinary retention measured by ultrasound and urodynamic study from baseline to 3 months post-operation or post transcutaneous stimulation
Change of urinary retention from baseline to 6 months post-operation or post transcutaneous stimulation | 6 months post surgery or post transcutaneous stimulation
  The change of volume of urinary retention measured by ultrasound and urodynamic study from baseline to 6 months post-operation or post transcutaneous stimulation
Change of urinary retention from baseline to 9 months post-operation or post transcutaneous stimulation | 9 months post surgery or post transcutaneous stimulation
  The change of volume of urinary retention measured by ultrasound and urodynamic study from baseline to 9 months post-operation or post transcutaneous stimulation
Change of urinary retention from baseline to 12 months post-operation or post transcutaneous stimulation | 12 months post surgery or post transcutaneous stimulation
  The change of volume of urinary retention measured by ultrasound and urodynamic study from baseline to 12 months post-operation or post transcutaneous stimulation
Change of urinary retention from baseline to 18 months post-operation or post transcutaneous stimulation | 18 months post surgery or post transcutaneous stimulation
  The change of volume of urinary retention measured by ultrasound and urodynamic study from baseline to 18 months post-operation or post transcutaneous stimulation
Change of urinary retention from baseline to 24 months post-operation or post transcutaneous stimulation | 24 months post surgery or post transcutaneous stimulation
  The change of volume of urinary retention measured by ultrasound and urodynamic study from baseline to 24 months post-operation or post transcutaneous stimulation
Change of MDS-UPDRS from baseline to immediately post-operation or post transcutaneous stimulation | Immediately post surgery or post transcutaneous stimulation
  The change of on-off rating of the Movement Disorders Society sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) from baseline to immediately post-operation or post transcutaneous stimulation
Change of MDS-UPDRS from baseline to 3 months post-operation or post transcutaneous stimulation | 3 months post surgery or post transcutaneous stimulation
  The change of on-off rating of the Movement Disorders Society sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) from baseline to 3 months post-operation or post transcutaneous stimulation
Change of MDS-UPDRS from baseline to 6 months post-operation or post transcutaneous stimulation | 6 months post surgery or post transcutaneous stimulation
  The change of on-off rating of the Movement Disorders Society sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) from baseline to 6 months post-operation or post transcutaneous stimulation
Change of MDS-UPDRS from baseline to 9 months post-operation or post transcutaneous stimulation | 9 months post surgery or post transcutaneous stimulation
  The change of on-off rating of the Movement Disorders Society sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) from baseline to 9 months post-operation or post transcutaneous stimulation
Change of MDS-UPDRS from baseline to 12 months post-operation or post transcutaneous stimulation | 12 months post surgery or post transcutaneous stimulation
  The change of on-off rating of the Movement Disorders Society sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) from baseline to 12 months post-operation or post transcutaneous stimulation
Change of MDS-UPDRS from baseline to 18 months post-operation or post transcutaneous stimulation | 18 months post surgery or post transcutaneous stimulation
  The change of on-off rating of the Movement Disorders Society sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) from baseline to 18 months post-operation or post transcutaneous stimulation
Change of MDS-UPDRS from baseline to 24 months post-operation or post transcutaneous stimulation | 24 months post surgery or post transcutaneous stimulation
  The change of on-off rating of the Movement Disorders Society sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) from baseline to 24 months post-operation or post transcutaneous stimulation
Change of UMSARS from baseline to 3 months post-operation or post transcutaneous stimulation | 3 months post surgery or post transcutaneous stimulation
  The change of on- off rating of the Unified Multiple System Atrophy Rating Scale (UMSARS) from baseline to 3 months post-operation or post transcutaneous stimulation
Change of UMSARS from baseline to 6 months post-operation or post transcutaneous stimulation | 6 months post surgery or post transcutaneous stimulation
  The change of on- off rating of the Unified Multiple System Atrophy Rating Scale (UMSARS) from baseline to 6 months post-operation or post transcutaneous stimulation
Change of UMSARS from baseline to 9 months post-operation or post transcutaneous stimulation | 9 months post surgery or post transcutaneous stimulation
  The change of on- off rating of the Unified Multiple System Atrophy Rating Scale (UMSARS) from baseline to 9 months post-operation or post transcutaneous stimulation
Change of UMSARS from baseline to 12 months post-operation or post transcutaneous stimulation | 12 months post surgery or post transcutaneous stimulation
  The change of on- off rating of the Unified Multiple System Atrophy Rating Scale (UMSARS) from baseline to 12 months post-operation or post transcutaneous stimulation
Change of UMSARS from baseline to 18 months post-operation or post transcutaneous stimulation | 18 months post surgery or post transcutaneous stimulation
  The change of on- off rating of the Unified Multiple System Atrophy Rating Scale (UMSARS) from baseline to 18 months post-operation or post transcutaneous stimulation
Change of UMSARS from baseline to 24 months post-operation or post transcutaneous stimulation | 24 months post surgery or post transcutaneous stimulation
  The change of on- off rating of the Unified Multiple System Atrophy Rating Scale (UMSARS) from baseline to 24 months post-operation or post transcutaneous stimulation
Change of UMSARS from baseline to immediately post-operation or post transcutaneous stimulation | Immediately post surgery or post transcutaneous stimulation
  The change of on- off rating of the Unified Multiple System Atrophy Rating Scale (UMSARS) from baseline to immediately post-operation or post transcutaneous stimulation
Change of lowest oxygen saturation from baseline to immediately post-operation or post transcutaneous stimulation | Immediately post surgery or post transcutaneous stimulation
  Change of lowest oxygen saturation measured by on-off polysomnography from baseline to immediately post-operation or post transcutaneous stimulation
Change of lowest oxygen saturation from baseline to 3 months post-operation or post transcutaneous stimulation | 3 months post surgery or post transcutaneous stimulation
  Change of lowest oxygen saturation measured by on-off polysomnography from baseline to 3 months post-operation or post transcutaneous stimulation
Change of lowest oxygen saturation from baseline to 6 months post-operation or post transcutaneous stimulation | 6 months post surgery or post transcutaneous stimulation
  Change of lowest oxygen saturation measured by on-off polysomnography from baseline to 6 months post-operation or post transcutaneous stimulation
Change of lowest oxygen saturation from baseline to 9 months post-operation or post transcutaneous stimulation | 9 months post surgery or post transcutaneous stimulation
  Change of lowest oxygen saturation measured by on-off polysomnography from baseline to 9 months post-operation or post transcutaneous stimulation
Change of lowest oxygen saturation from baseline to 12 months post-operation or post transcutaneous stimulation | 12 months post surgery or post transcutaneous stimulation
  Change of lowest oxygen saturation measured by on-off polysomnography from baseline to 12 months post-operation or post transcutaneous stimulation
Change of lowest oxygen saturation from baseline to 18 months post-operation or post transcutaneous stimulation | 18 months post surgery or post transcutaneous stimulation
  Change of lowest oxygen saturation measured by on-off polysomnography from baseline to 18 months post-operation or post transcutaneous stimulation
Change of lowest oxygen saturation from baseline to 24 months post-operation or post transcutaneous stimulation | 24 months post surgery or post transcutaneous stimulation
  Change of lowest oxygen saturation measured by on-off polysomnography from baseline to 24 months post-operation or post transcutaneous stimulation
Change of mean oxygen saturation from baseline to immediately post-operation or post transcutaneous stimulation | Immediately post surgery or post transcutaneous stimulation
  Change of mean oxygen saturation measured by on-off polysomnography from baseline to immediately post-operation or post transcutaneous stimulation
Change of mean oxygen saturation from baseline to 3 months post-operation or post transcutaneous stimulation | 3 months post surgery or post transcutaneous stimulation
  Change of mean oxygen saturation measured by on-off polysomnography from baseline to 3 months post-operation or post transcutaneous stimulation
Change of mean oxygen saturation from baseline to 6 months post-operation or post transcutaneous stimulation | 6 months post surgery or post transcutaneous stimulation
  Change of mean oxygen saturation measured by on-off polysomnography from baseline to 6 months post-operation or post transcutaneous stimulation
Change of mean oxygen saturation from baseline to 9 months post-operation or post transcutaneous stimulation | 9 months post surgery or post transcutaneous stimulation
  Change of mean oxygen saturation measured by on-off polysomnography from baseline to 9 months post-operation or post transcutaneous stimulation
Change of mean oxygen saturation from baseline to 12 months post-operation or post transcutaneous stimulation | 12 months post surgery or post transcutaneous stimulation
  Change of mean oxygen saturation measured by on-off polysomnography from baseline to 12 months post-operation or post transcutaneous stimulation
Change of mean oxygen saturation from baseline to 18 months post-operation or post transcutaneous stimulation | 18 months post surgery or post transcutaneous stimulation
  Change of mean oxygen saturation measured by on-off polysomnography from baseline to 18 months post-operation or post transcutaneous stimulation
Change of mean oxygen saturation from baseline to 24 months post-operation or post transcutaneous stimulation | 24 months post surgery or post transcutaneous stimulation
  Change of mean oxygen saturation measured by on-off polysomnography from baseline to 24 months post-operation or post transcutaneous stimulation
Change of SCOPA-AUT from baseline to immediately post-operation or post transcutaneous stimulation | Immediately post surgery or post transcutaneous stimulation
  Change of scales for outcomes in Parkinson's disease - autonomic dysfunction from baseline to immediately post-operation or post transcutaneous stimulation
Change of SCOPA-AUT from baseline to 3 months post-operation or post transcutaneous stimulation | 3 months post surgery or post transcutaneous stimulation
  Change of scales for outcomes in Parkinson's disease - autonomic dysfunction from baseline to 3 months post-operation or post transcutaneous stimulation
Change of SCOPA-AUT from baseline to 6 months post-operation or post transcutaneous stimulation | 6 months post surgery or post transcutaneous stimulation
  Change of scales for outcomes in Parkinson's disease - autonomic dysfunction from baseline to 6 months post-operation or post transcutaneous stimulation
Change of SCOPA-AUT from baseline to 9 months post-operation or post transcutaneous stimulation | 9 months post surgery or post transcutaneous stimulation
  Change of scales for outcomes in Parkinson's disease - autonomic dysfunction from baseline to 9 months post-operation or post transcutaneous stimulation
Change of SCOPA-AUT from baseline to 12 months post-operation or post transcutaneous stimulation | 12 months post surgery or post transcutaneous stimulation
  Change of scales for outcomes in Parkinson's disease - autonomic dysfunction from baseline to 12 months post-operation or post transcutaneous stimulation
Change of SCOPA-AUT from baseline to 18 months post-operation or post transcutaneous stimulation | 18 months post surgery or post transcutaneous stimulation
  Change of scales for outcomes in Parkinson's disease - autonomic dysfunction from baseline to 18 months post-operation or post transcutaneous stimulation
Change of SCOPA-AUT from baseline to 24 months post-operation or post transcutaneous stimulation | 24 months post surgery or post transcutaneous stimulation
  Change of scales for outcomes in Parkinson's disease - autonomic dysfunction from baseline to 24 months post-operation or post transcutaneous stimulation
Change of delta cerebral artery velocity from baseline to immediately post-operation or post transcutaneous stimulation | Immediately post surgery or post transcutaneous stimulation
  Change of on-off delta cerebral artery velocity from baseline to immediately post-operation or post transcutaneous stimulation. Delta cerebral artery velocity equals cerebral artery velocity of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes.
Change of delta cerebral artery velocity from baseline to 3 months post-operation or post transcutaneous stimulation | 3 months post surgery or post transcutaneous stimulation
  Change of on-off delta cerebral artery velocity from baseline to 3 months post-operation or post transcutaneous stimulation. Delta cerebral artery velocity equals cerebral artery velocity of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes.
Change of delta cerebral artery velocity from baseline to 6 months post-operation or post transcutaneous stimulation | 6 months post surgery or post transcutaneous stimulation
  Change of on-off delta cerebral artery velocity from baseline to 6 months post-operation or post transcutaneous stimulation. Delta cerebral artery velocity equals cerebral artery velocity of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes.
Change of delta cerebral artery velocity from baseline to 9 months post-operation or post transcutaneous stimulation | 9 months post surgery or post transcutaneous stimulation
  Change of on-off delta cerebral artery velocity from baseline to 9 months post-operation or post transcutaneous stimulation. Delta cerebral artery velocity equals cerebral artery velocity of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes.
Change of delta cerebral artery velocity from baseline to 12 months post-operation or post transcutaneous stimulation | 12 months post surgery or post transcutaneous stimulation
  Change of on-off delta cerebral artery velocity from baseline to 12 months post-operation or post transcutaneous stimulation. Delta cerebral artery velocity equals cerebral artery velocity of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes.
Change of delta cerebral artery velocity from baseline to 18 months post-operation or post transcutaneous stimulation | 18 months post surgery or post transcutaneous stimulation
  Change of on-off delta cerebral artery velocity from baseline to 18 months post-operation or post transcutaneous stimulation. Delta cerebral artery velocity equals cerebral artery velocity of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes.
Change of delta cerebral artery velocity from baseline to 24 months post-operation or post transcutaneous stimulation | 24 months post surgery or post transcutaneous stimulation
  Change of on-off delta cerebral artery velocity from baseline to 24 months post-operation or post transcutaneous stimulation. Delta cerebral artery velocity equals cerebral artery velocity of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes.
Change of TUG from baseline to immediately post-operation or post transcutaneous stimulation | Immediately post surgery or post transcutaneous stimulation
  Change of on-off timed up and go from baseline to immediately post-operation or post transcutaneous stimulation
Change of TUG from baseline to 3 months post-operation or post transcutaneous stimulation | 3 months post surgery or post transcutaneous stimulation
  Change of on-off timed up and go from baseline to 3 months post-operation or post transcutaneous stimulation
Change of TUG from baseline to 6 months post-operation or post transcutaneous stimulation | 6 months post surgery or post transcutaneous stimulation
  Change of on-off timed up and go from baseline to 6 months post-operation or post transcutaneous stimulation
Change of TUG from baseline to 9 months post-operation or post transcutaneous stimulation | 9 months post surgery or post transcutaneous stimulation
  Change of on-off timed up and go from baseline to 9 months post-operation or post transcutaneous stimulation
Change of TUG from baseline to 12 months post-operation or post transcutaneous stimulation | 12 months post surgery or post transcutaneous stimulation
  Change of on-off timed up and go from baseline to 12 months post-operation or post transcutaneous stimulation
Change of TUG from baseline to 18 months post-operation or post transcutaneous stimulation | 18 months post surgery or post transcutaneous stimulation
  Change of on-off timed up and go from baseline to 18 months post-operation or post transcutaneous stimulation
Change of TUG from baseline to 24 months post-operation or post transcutaneous stimulation | 24 months post surgery or post transcutaneous stimulation
  Change of on-off timed up and go from baseline to 24 months post-operation or post transcutaneous stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology and Institute of Neurology, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai 200025 Recruiting, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No